CLINICAL TRIAL: NCT02100150
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of NNZ-2566 in the Acute Treatment of Adolescents and Adults With Mild Traumatic Brain Injury (mTBI)
Brief Title: A Safety and Efficacy Study of NNZ-2566 in Patients With Mild Traumatic Brain Injury (mTBI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neu-2566-TBI-003
Record Dates: First submitted 2014-03-19; First posted 2014-03-31 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Concussion
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — trofinetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNZ-2566 (Experimental): Glycyl-L-2-Methylpropyl-L-Glutamic Acid
  Interventions: Drug: NNZ-2566
- Placebo (strawberry flavored solution) (Placebo Comparator): Strawberry flavored solution and water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2566 — Glycyl-L-2-Methylpropyl-L-Glutamic Acid (NNZ-2566) supplied as a lyophilized powder (3g in 30 milliliter vials) for reconstitution with strawberry flavored solution 0.5% v/v in Water for Injection.
  Arms: NNZ-2566
Drug: Placebo — Strawberry flavored solution 0.5% v/v in Water for Injection
  Other Names: Strawberry flavored solution
  Arms: Placebo (strawberry flavored solution)

SUMMARY:
The purpose of this study is to determine whether NNZ-2566 is safe and well tolerated in the treatment of mTBI in adolescents and adults.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is an injury to the head caused by an external trauma that can lead to brain cell death, inflammation, edema, hemorrhage, and disruption of normal brain cell function. mTBI frequently results in persistent functional impairment including problems with cognitive function, memory, mood, and other personality disorders.

There are currently no drugs available to reduce the brain damage or sequelae that result from TBI. Clearly, a safe and effective treatment for concussion injury and all forms of TBI would be an important development for military personnel as well as the general population.

This study will investigate the safety and tolerability of treatment with oral administration of NNZ-2566 at 35 mg/kg or 70 mg/kg BID in adolescents and adults with mTBI. The study also will also investigate measures of efficacy during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of mTBI resulting from an injury that meets the following criteria:

   1. Occurred within 24 hours of Screening and was associated with a clear mechanism of injury and an alteration of consciousness (e.g., confusion, feeling dazed, or "seeing stars")
   2. Was associated with a GCS score of 13-15
   3. Was associated with 1 or more of the following signs and symptoms, as determined by a qualified clinician:

   i. Headache ii. Loss of consciousness iii. Post traumatic amnesia iv. Retrograde amnesia v. Difficulty concentrating vi. Balance problems vii. Dizziness viii. Visual problems ix. Personality changes x. Fatigue xi. Sensitivity to light/noise xii. Numbness xiii. Nausea xiv. Vomiting d. Current symptoms associated with the mTBI are causing clinically significant impairment
2. Subject is 16 to 55 years old.
3. Subject has a CGI-S score of ≥3 at Screening
4. Subject has an RPQ-3 score of ≥3 at Screening
5. Subjects who are taking psychotropic medications must have been receiving a stable regimen (i.e., same dosage and regimen) for at least 4 weeks prior to Screening. For the purposes of this protocol, psychotropic medications are defined as medications that are prescribed for intended CNS benefits. Medications for headache are permissible, as needed, according to approved prescribing information.
6. Women of child-bearing potential must have a negative urine pregnancy test at Screening. Men and women must agree to use a contraceptive method with <1% success rate (e.g., oral contraceptive, injectable progestogen, levonorgestrel implant, estrogenic vaginal ring, percutaneous contraceptive patch, intrauterine device [IUD], surgical sterilization, or double barrier method [i.e., condom with diaphragm or spermicidal agent]).

Exclusion Criteria:

Subjects are ineligible for the study if they meet any of the following exclusion criteria:

1. Subject has a history of brain surgery or prior severe TBI (based on a previously documented GCS score of ≤8).
2. Subject has a history of seizure disorder or has experienced seizures in the 24 hours preceding Screening. Note: Isolated febrile seizures during early childhood are not exclusionary.
3. Subject has a history of diabetes mellitus requiring pharmacotherapy within the preceding 12 months.
4. Subject has a history of hypothyroidism within the 3 years preceding Screening that currently requires or did require pharmacotherapy.
5. Subject has regularly used more than 1 of the following psychoactive medications in the 4 weeks preceding Screening: methylphenidate, dextroamphetamine, mixed amphetamine salts, amantadine, memantine, cholinesterase inhibitors, modafinil, or armodafinil.
6. Subject has a history of substance abuse or dependence, other than nicotine dependence, within the 3 months preceding Screening.
7. Subject has signs/symptoms of acute impairment due to alcohol use.
8. Subject has used anti-epileptic medications in the 4 weeks preceding Screening.
9. Subject has used bromocryptine, levodopa, ropinirole, or pramipexole in the 4 weeks preceding Screening.
10. Subject has a history of a major psychiatric disorder (including major depression, a clinically significant anxiety disorder, or a psychotic disorder) that is associated with significant clinical impairment within the preceding 6 months.
11. In the Investigator's opinion, the subject poses a current homicidal or serious suicidal risk, and/or has made a suicide attempt within the 6 months preceding Screening.
12. Subject has a neurological disorder other than mTBI (e.g., Parkinson's disease, stroke, multiple sclerosis, dementia, delirium, infectious encephalopathy) that has required treatment within the 6 months preceding Screening.
13. Subject has a history of, or current, cerebrovascular disease.
14. Subject has a history of, or current, malignancy.
15. Subject has an unstable medical disorder that may pose a safety concern or interfere with the accurate assessment of safety or efficacy.
16. Subject has laboratory values at Screening deemed to be clinically significant by the Investigator.
17. Subject has an average QT interval corrected using Fridericia's formula (QTcF) >450 msec at Screening or any ECG abnormality that may pose a potential safety concern.
18. Subject has a history of risk factors for torsade de pointes (e.g., heart failure, clinically significant hypokalemia, a serum potassium value at Screening of <3.0 mmol/L, or a family history of long QT syndrome).
19. Subject has a history of QT/QTcF prolongation previously or currently controlled with medication, in which normal QT/QTcF intervals could or can only be achieved with medication.
20. Subject has participated in another clinical treatment study within the 4 weeks preceding Screening.
21. Subject is unable to provide informed consent (where deemed cognitively able by standard assessments) or informed consent cannot be obtained from a legally authorized individual (e.g., spouse, or in the instance of minors, a parent).
22. Subject is pregnant or nursing.
23. Subject was previously enrolled in this study.
24. Subject has an allergy to strawberries.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cognitive Function - Automated Neuropsychological Assessment Metrics (ANAM) | Through to Day 28
  The ANAM is a library of computerized tests that measures 6 cognitive domains believed to be most highly impacted by mTBI: simple reaction time, procedural reaction time, learning, working memory, delayed memory, and spatial memory.
  Only selected subtests of the ANAM will be performed during this study, as follows:
  * Code substitution - learning, simple reaction time, procedural reaction time, code substitution.
  * Simple reaction time and procedural reaction time.
General Clinical Status - Clinical Global Impression of Severity and Improvement (CGI-S, CGI-I) | Through to Day 28
  The CGI-S is an assessment that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis.
Post-Injury Symptoms | Through to Day 28
  Residual self-reported symptoms associated with mTBI will be assessed using the Post-Concussion Symptom Scale (PCSS).
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) is used to measure the presence and severity of post-concussion syndrome, which addresses a set of somatic, cognitive, and emotional symptoms following TBI.
Postural Stability | Through to Day 28.
  Postural sway will be analysed using the Sway Balance Application. Sway Balance will be measured using the Balance Error Scoring System (BESS). Pupil size and dynamics as well as the associated neurological pupillary index (NPi) will be measured using a handheld, infrared, digital pupillometer.
  An Accommodation/Convergence test will be performed. Convergence is the inward rotational ability of the eye. Accommodation is the ability of the eye to maintain focus as the distance changes.
Psychological Sequelae | Through to Day 28
  Anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS).
  Post-traumatic stress disorder will be measured by the Post-Traumatic Stress Disorder Checklist-Specific (PCL-S).
Change in subject's readiness and fitness to return to work as measured by the Return-to-Duty Assessment | Day 3 to 28
  The Return-to-Duty Assessment is a standardized protocol to determine a subject's readiness or fitness to return to duty (yes/no). Once the subject has been cleared to return to duty, this assessment is no longer applicable for that subject.
Residual Functional Disability | Day 28
  Residual Functional Ability will be measured by the Sheehan Disability Scale (SDS) which measures the extent to which 3 major sectors in the subject's life are impaired by an illness or disorder.

SECONDARY OUTCOMES:
Safety | Screening through to Day 28 or the final study visit, whichever comes later
  Incidence of adverse events (AE), including Serious adverse events (SAE), will be evaluated between the two NNZ-2566 doses and placebo. Incidence of AEs and SAEs will be evaluated from randomized dosing through to Day 28 or the final study visit, whichever comes later.
Pharmacodynamic Measurements of Protein Biomarkers and micro-RNA | Screening through to Day 3
  A blood sample will be obtained to measure levels of protein biomarkers (SBDP150, S100, GFAP, and UCH-L1) that are derived from the cytosol of neurons, astrocytes, axons; micro-RNA (mi-RNA) levels will also be measured. This blood sample will be obtained at Screening, and on Days 1, 2, and 3.
Pharmacokinetic (PK) Measurements - maximum observed concentration (Cmax), trough concentration (Cmin),and area under the concentration-time curve (AUC) at steady-state | Day 3 and Day 7
  The following pharmacokinetic measures will be calculated from NNZ-2566 concentrations in whole blood: Cmax, Cmin, and AUC at steady-state.
  A PK blood sample (2 x 2 mL) will be collected on Day 3 at approximately 2 to 4 hours after administration of study drug, and on Day 7 at pre-dose and approximately 4 hours after administration of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley R Cole, Ph.D, Principal Investigator — Fort Bragg; Kurt Denninghoff, MD, Principal Investigator — University of Arizona; Alex Hishaw, MD, Principal Investigator — University of Arizona; Brian O'Neil, MD, Principal Investigator — Detroit Receiving Hospital
Locations (1):
- Fort Bragg, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided